CLINICAL TRIAL: NCT05206578
Title: To Evaluate the Efficacy and Safety of Combination Therapy of AGT and AGZ Versus Monotherapy of AGT in Patients With Primary Hypercholesterolemia
Brief Title: Study to Evaluate the Efficacy and Safety in Patients With Primary Hypercholesterolemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG1901 P3
Record Dates: First submitted 2022-01-12; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Primary Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AGT2, AGZ (Experimental)
  Interventions: Drug: AGT2, AGZ
- AGT2 (Active Comparator)
  Interventions: Drug: AGT2
- AGT4, AGZ (Experimental)
  Interventions: Drug: AGT4, AGZ
- AGT4 (Active Comparator)
  Interventions: Drug: AGT4

INTERVENTIONS:
Drug: AGT2, AGZ — Tablet, q.d.
  Arms: AGT2, AGZ
Drug: AGT2 — Tablet, q.d.
  Arms: AGT2
Drug: AGT4, AGZ — Tablet, q.d.
  Arms: AGT4, AGZ
Drug: AGT4 — Tablet, q.d.
  Arms: AGT4

SUMMARY:
To Evaluate the Efficacy and Safety of Combination Therapy of AGT and AGZ Versus Monotherapy of AGT in Patients With Primary Hypercholesterolemia.

DETAILED DESCRIPTION:
A Multi-center, Randomized, Double-blinded, Active-controlled, Factorial Design Phase 3 Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary hypercholesterolemia

Exclusion Criteria:

* The subject not meet the specified LDL-C level

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-07-07 (Estimated); Study Completion 2022-09-08 (Estimated)

PRIMARY OUTCOMES:
% change in LDL-C level from baseline at Week 8 | Week 8
  change in LDL-C level

SECONDARY OUTCOMES:
Change in LDL-C level from baseline at Week 4 | Week 4
  change in LDL-C level

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei severance Hospital, Seoul, South Korea